CLINICAL TRIAL: NCT01772160
Title: Population Based Surveillance to Estimate the Burden of Herpes Zoster and Post-herpetic Neuralgia in Italy
Brief Title: Study to Estimate the Burden of Herpes Zoster (HZ) and Post-herpetic Neuralgia (PHN) in Italy
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116208
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Herpes Zoster; Herpes Zoster Vaccine
Keywords: Adults; Italy; Herpes Zoster; Complications; Quality of life; Surveillance; Burden; Cost; Incidence
MeSH Terms: conditions — Herpes Zoster | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Herpes Zoster Group: Male or female subjects aged 50 years or above, presenting with a herpes zoster (HZ) episode.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — HZ/PHN booklet, HZ/PHN file and logbook. HZ/PHN booklet will be completed by the patient and the HZ/PHN file and logbook will be completed by the participating general practitioner.

SUMMARY:
The purpose of this study is to collect data on the incidence, complications, economic burden and impact on the quality of life in adults aged ≥ 50 years with HZ disease in Italy.

DETAILED DESCRIPTION:
The surveillance/recruitment period will take approximately 2 years and once the enrolment of HZ patients has ended, the study will continue for a maximum of 9 months to allow for completion of the follow-up of potential PHN cases.

The data will be captured at protocol specified time-points based on the time of enrolment of each subject.

ELIGIBILITY:
Inclusion Criteria:

* A male or female ≥ 50 years of age at the time of study enrolment presenting with acute HZ.
* HZ diagnosis for this HZ episode:

  * Is his/her first outpatient diagnosis (i.e. initial consultation), OR
  * Took place at another site/centre (e.g. emergency room or Dermatologist/Specialist practice) provided the HZ diagnosis is not more than 7 days before the initial visit for the present study (i.e. secondary consultation).
* Written informed consent obtained from the patient.
* Ability to comply with study procedures.

Exclusion Criteria:

• Patient participating in another clinical study (participation in another observational, non-interventional trial is allowed).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population, male or female aged ≥ 50 years of age presenting with a HZ episode.
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2013-02-26 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (35):
- Italy (35):
  - GSK Investigational Site, Cavallino (LE), Apulia
  - GSK Investigational Site, Copertino (LE), Apulia
  - GSK Investigational Site, Cutrofiano (LE), Apulia
  - GSK Investigational Site, Galatina (LE), Apulia
  - GSK Investigational Site, Montesano S. (LE), Apulia
  - GSK Investigational Site, Parabita (LE), Apulia
  - GSK Investigational Site, Specchia (LE), Apulia
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Angera (VA), Lombardy
  - GSK Investigational Site, Arcisate (VA), Lombardy
  - GSK Investigational Site, Comerio (VA), Lombardy
  - GSK Investigational Site, Fagnano Olona (VA), Lombardy
  - GSK Investigational Site, Ghirla Valganna (VA), Lombardy
  - GSK Investigational Site, Induno Olona (VA), Lombardy
  - GSK Investigational Site, Sesto Calende (VA), Lombardy
  - GSK Investigational Site, Solbiate Olona (VA), Lombardy
  - GSK Investigational Site, Varese, Lombardy
  - GSK Investigational Site, Alessandria, Piedmont
  - GSK Investigational Site, Frugarolo (AL), Piedmont
  - GSK Investigational Site, Oviglio (AL), Piedmont
  - GSK Investigational Site, Sale (AL), Piedmont
  - GSK Investigational Site, Villalvernia (AL), Piedmont
  - GSK Investigational Site, Arcidosso (GR), Tuscany
  - GSK Investigational Site, Arezzo, Tuscany
  - GSK Investigational Site, Civitella Paganico (GR), Tuscany
  - GSK Investigational Site, Follonica (GR), Tuscany
  - GSK Investigational Site, Grosseto, Tuscany
  - GSK Investigational Site, Lucignano (AR), Tuscany
  - GSK Investigational Site, Orbetello (GR), Tuscany
  - GSK Investigational Site, Sassofortino (GR), Tuscany
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Ripa (PG), Umbria
  - GSK Investigational Site, Alessano (LE)
  - GSK Investigational Site, Rome

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20346

REFERENCES:
- [Background] Salvetti A, Ferrari V, Garofalo R, Gazzaniga P, Guerroni A, Metrucci A, Sessa A, Severi ML, Nati G, Ruggeri M, Rossi A, Cappellari L, Gopala K, Tosatto R, Simone B. Incidence of herpes zoster and postherpetic neuralgia in Italian adults aged >/=50 years: A prospective study. Prev Med Rep. 2019 Apr 24;14:100882. doi: 10.1016/j.pmedr.2019.100882. eCollection 2019 Jun. PMID 31193254
- [Derived] Matthews S, De Maria A, Passamonti M, Ristori G, Loiacono I, Puggina A, Curran D. The Economic Burden and Impact on Quality of Life of Herpes Zoster and Postherpetic Neuralgia in Individuals Aged 50 Years or Older in Italy. Open Forum Infect Dis. 2019 Jan 12;6(2):ofz007. doi: 10.1093/ofid/ofz007. eCollection 2019 Feb. PMID 30793003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 395 subjects originally enrolled in this study, 1 subject was excluded due to protocol violation, hence only 394 were included in the Total Cohort.
Period: Overall Study
Arm/Group | Herpes Zoster Group
Started | 394
Completed | 346
Not Completed | 48
Not completed — Death | 3
Not completed — Eligibility criteria not fulfilled | 3
Not completed — Consent withdrawal | 3
Not completed — Migrated / moved from the study area | 4
Not completed — Lost to Follow-up | 30
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 394
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238
  Male | 156
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Incidence Rate of Herpes Zoster (HZ) Cases, by Age and Gender
Description: A case of HZ was defined as new unilateral pain (broadly defined to include allodynia and pruritus) accompanied by unilateral rash and no alternative diagnosis. Age ranges were 50-54, 55-59, 60-64, 65-69, 70-74, 75-79 and greater than or equal to (≥) 80 years. The incidence rate was expressed as the number of HZ cases per (/) 1000 person-years.
Time Frame: Day 0 to 2 years
Population: The analysis was performed on the HZ cases occurring in the total population covered by the participating general practitioners (GPs).
Measure: Mean (95% Confidence Interval); unit: Number of HZ cases/1000 person-years
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 721
Number of HZ cases/1000 person-years
  Female, 50-54: number analyzed (Participants) | 49
  Female, 50-54 | 5.19 [3.84 to 6.86]
  Female, 55-59: number analyzed (Participants) | 56
  Female, 55-59 | 6.29 [4.75 to 8.17]
  Female, 60-64: number analyzed (Participants) | 39
  Female, 60-64 | 5.00 [3.55 to 6.83]
  Female, 65-69: number analyzed (Participants) | 74
  Female, 65-69 | 9.19 [7.22 to 11.54]
  Female, 70-74: number analyzed (Participants) | 54
  Female, 70-74 | 7.51 [5.64 to 9.79]
  Female, 75-79: number analyzed (Participants) | 71
  Female, 75-79 | 10.72 [8.37 to 13.52]
  Female, ≥ 80: number analyzed (Participants) | 92
  Female, ≥ 80 | 7.06 [5.69 to 8.65]
  Male, 50-54: number analyzed (Participants) | 15
  Male, 50-54 | 1.71 [0.96 to 2.82]
  Male, 55-59: number analyzed (Participants) | 23
  Male, 55-59 | 2.91 [1.85 to 4.37]
  Male, 60-64: number analyzed (Participants) | 32
  Male, 60-64 | 4.35 [2.98 to 6.15]
  Male, 65-69: number analyzed (Participants) | 62
  Male, 65-69 | 8.95 [6.86 to 11.47]
  Male, 70-74: number analyzed (Participants) | 56
  Male, 70-74 | 9.33 [7.05 to 12.12]
  Male, 75-79: number analyzed (Participants) | 39
  Male, 75-79 | 7.18 [5.10 to 9.81]
  Male, ≥ 80: number analyzed (Participants) | 59
  Male, ≥ 80 | 7.20 [5.48 to 9.29]
  Overall incidence of HZ cases | 6.46 [5.99 to 6.95]

2. Secondary Outcome: Percentage of Postherpetic Neuralgia (PHN) Cases Among HZ, Overall
Description: PHN persistence refers to pain occurring or persisting from Day 90 to Day 270 after the rash onset. PHN was assessed via the Zoster Pain Inventory (ZBPI) questionnaire, which includes four pain severity items (worst, least, average, present pain) and seven pain interference items which assess general activity, mood, walking ability, work, relations with others, sleep and enjoyment of life. All of the items are rated on an 11-point Likert scale (0-10). For the severity items, 0 = 'no pain' and 10 = 'pain as bad as you can imagine', whereas for the interference items, 0 = 'does not interfere' and 10 = 'completely interferes'.
Time Frame: At Day 90, 180 and 270 after onset of HZ
Population: The analysis was performed on the HZ cases (with completed questionnaires up to Day 270) occurring in the According-To-Protocol cohort (ATP) which included all evaluable patients (i.e. those who met all eligibility criteria and complied with the study procedures defined in the protocol).
Measure: Number (95% Confidence Interval); unit: Percentage of PHN cases
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 343
Percentage of PHN cases
  Overall PHN cases, Day 90 | 11.66 [8.46 to 15.54]
  Overall PHN cases, Day 180: number analyzed (Participants) | 14
  Overall PHN cases, Day 180 | 42.86 [17.66 to 71.14]
  Overall PHN cases, Day 270: number analyzed (Participants) | 4
  Overall PHN cases, Day 270 | 75.00 [19.41 to 99.37]

3. Secondary Outcome: General Medical History of Cases With HZ, Overall
Description: General medical history focused on characteristics such as patient pre-existing condition and diseases (local trauma, diabetes mellitus, liver disease, alcoholism, renal failure/dialysis, emotional problems, stress or depression, blood malignancy, solid malignancy, hematopoetic cell/ bone marrow transplant, solid organ transplantation, HIV infection, hepatitis C under active therapy, autoimmune disease active and under therapy, other).
Time Frame: Between Day 0 and Day 270.
Population: The analysis was performed on the HZ cases occurring in the According-To-Protocol cohort (ATP) which included all evaluable patients (i.e. those who met all eligibility criteria and complied with the study procedures defined in the protocol).
Measure: Number; unit: Percentage of HZ cases
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 391
Percentage of HZ cases
  Pre-existing condition, Yes | 32.74
  Pre-existing condition, No | 67.26
  Pre-existing condition, Missing Confirmed | 0.00
  Local Trauma | 3.91
  Diabetes mellitus | 35.94
  Liver disease | 4.69
  Alcoholism | 2.34
  Renal failure/dialysis | 7.03
  Emotional problems, stress or depression | 32.03
  Blood malignancy | 0.78
  Solid malignancy | 3.91
  Hematopoetic cell/ bone marrow transplant | 0.00
  Solid organ transplantation | 0.78
  HIV infection | 0.78
  Hepatitis C under active therapy | 0.78
  Autoimmune disease active and under therapy | 5.47
  Other | 25.00

4. Secondary Outcome: Other General Medical History Characteristics for HZ Cases, Overall
Description: Other general medical history characteristics referred to arterial problems, cerebral problems, gastric problems, gastric problems, prostate problems (arterial hypertension and allergic rhinitis, arterial hypertension and pacemaker, arteriopathy and past nun-Hodgkin lymphoma, atrial fibrillation, bronchopathy, cerebral thrombosis, cholecyst, chronic cerebral ischemia, chronic leukemia, chronic obstructive pulmonary disease, epilepsy, gastric lymphoma, gastropathy, hypertension, hypertension and hypothyroidism after surgery, hypertension dyslipidemia and hyperthyroidism, hypothyroidism hypertension, polycythaemia, polycythaemia from 10 years, prostate neoplasm, prostate oral anticoagulant therapy cardiopathy, prostatic cancer, right feet arthralgia, thrombocytopenia, vasculopathy chronic brain).
Time Frame: Between Day 0 and Day 270.
Population: as for outcome 3
Measure: Number; unit: Percentage of HZ cases
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 32
Percentage of HZ cases
  Arterial hypertension and allergic rhinitis | 3.13
  Arterial hypertension and pacemaker | 3.13
  Arteriopathy and past non-Hodgkin lymphoma | 3.13
  Atrial fibrillation | 3.13
  Bronchopathy | 3.13
  Cerebral thrombosis | 3.13
  Cholecyst | 3.13
  Chronic cerebral ischemia | 3.13
  Chronic leukemia | 3.13
  Chronic obstructive pulmonary disease | 3.13
  Epilepsy | 3.13
  Gastric lymphoma | 3.13
  Gastropathy | 3.13
  Hypertension | 25.00
  Hypertension and hypothyroidism after surgery | 3.13
  Hypertension dyslipidemia and hyperthyroidism | 3.13
  Hypothyroidism hypertension | 3.13
  Polycythaemia | 3.13
  Polycythaemia from 10 years | 3.13
  Prostate neoplasm | 3.13
  Prostate oral anticoagulant therapy cardiopathy | 3.13
  Prostatic cancer | 3.13
  Right feet arthralgia | 3.13
  Thrombocytopenia | 3.13
  Vasculopathy chronic brain | 3.13

5. Secondary Outcome: Clinical Information of Cases With HZ, Overall
Description: Clinical information of HZ cases referred to experience of any symptoms before rash, actual symptoms before rash (SBR), any complications at initial visit.
Time Frame: Between Day 0 and Day 270
Population: as for outcome 3
Measure: Number; unit: Percentage of HZ cases
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 391
Percentage of HZ cases
  Any symptoms before rash, Yes | 73.66
  Any symptoms before rash, No | 26.34
  SBR, Prodromal pain | 82.64
  SBR, Fever | 5.90
  SBR, Malaise | 29.17
  SBR, Other:Ailment to the touch | 0.35
  SBR, Other:Burning sensation | 3.13
  SBR, Other:Dysesthesia | 0.35
  SBR, Other:Fever sensation | 0.35
  SBR, Other:Itching feeling of internal heat | 0.35
  SBR, Other:Itching | 6.25
  SBR, Other:Paresthesia | 0.35
  SBR, Other:Pain in right eyelid | 0.35
  SBR, Other:Pain in upper arms | 0.35
  SBR, Other:Sweating | 0.00
  Any complications at initial visit, Yes | 16.62
  Any complications at initial visit, No | 83.38

6. Secondary Outcome: Complications Related to HZ Cases, Overall
Description: HZ related complications refer to cutaneous complications (Varicella Zoster Virus [VZV] dissemination, Bacterial superinfection), ocular (Loss of corneal sensation, Keratitis, Scleritis, Uveitis, Iridocyclitis), neurological (Meningo-encephalitis, Cranial nerve palsies, Peripheral nerve palsies, Ramsay-Hunt syndrome, Persistent HZ-related Pain), visceral [Neural extension of VZV infection (bronchitis, esophagitis,cystitis), VZV dissemination (pneumonia, arthritis, hepatitis] and other.
Time Frame: Between Day 0 and Day 270
Population: as for outcome 3
Measure: Number; unit: Percentage of HZ complications
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 65
Percentage of HZ complications
  VZV dissemination | 44.62
  Bacterial superinfection | 7.69
  Loss of corneal sensation | 0.00
  Keratitis | 10.77
  Scleritis | 0.00
  Uveitis | 4.62
  Iridocyclitis | 1.54
  Meningo-encephalitis | 0.00
  Cranial nerve palsies | 3.08
  Peripheral nerve palsies | 0.00
  Ramsay-Hunt syndrome | 0.00
  Persistent HZ-related Pain | 64.62
  Neural extension of VZV infection | 0.00
  Pneumonia, arthritis, hepatitis | 1.54
  Other | 7.69

7. Secondary Outcome: Other Complications Related to HZ Cases, Overall
Description: HZ related other complications refer to axillary lympagenopathy, burning sensation, hypoacusis, itching and rectum pain.
Time Frame: Between Day 0 and Day 270
Population: as for outcome 3
Measure: Number; unit: Percentage of HZ complications
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 5
Percentage of HZ complications
  Axillary lymphadenopathy | 20.00
  Burning sensation | 20.00
  Hypoacusis | 20.00
  Itching | 20.00
  Rectum pain | 20.00

8. Secondary Outcome: Direct Medical Costs, Direct Non-medical Costs and Indirect Costs
Description: Cost data related to HZ included medication, procedures and referral to hospital/specialist for direct medical costs, transport for direct non-medical costs and missed time from work, sick certificate for the indirect costs.
Time Frame: Up to Day 90
Population: The analysis was performed on the HZ subjects from the According-To-Protocol cohort (ATP) which included all evaluable patients (i.e. those who met all eligibility criteria and complied with the study procedures defined in the protocol).
Measure: Mean (Standard Deviation); unit: Euro
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 391
Euro
  Direct Medical Cost | 189 (377)
  Productivity Loss - Subject: number analyzed (Participants) | 17
  Productivity Loss - Subject | 2124 (1965)
  Productivity Loss - Caregiver: number analyzed (Participants) | 12
  Productivity Loss - Caregiver | 82 (105)
  Transport | 13 (54)
  Overall | 297 (730)

9. Secondary Outcome: Worst Pain Assessment in HZ Subjects
Description: The ZBPI is an assessment tool in the form of a questionnaire completed by the patient that is specifically designed to assess HZ-associated pain and discomfort. the ZBPI includes four pain severity items (worst, least, average, present pain) and seven pain interference items which assess general activity, mood, walking ability, work, relations with others, sleep and enjoyment of life. All of the items are rated on an 11-point Likert scale (0-10). For the severity items, 0 = 'no pain' and 10 = 'pain as bad as you can imagine', whereas for the interference items, 0 = 'does not interfere' and 10 = 'completely interferes'. Note: The Day 90 window included assessments between Day 83 and Day 97 relative to day of rash onset.
Time Frame: At Day 90
Population: The analysis was performed on the According-To-Protocol cohort (ATP) which included all evaluable patients (i.e. those who met all eligibility criteria and complied with the study procedures defined in the protocol).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 391
Scores on a scale | 0.7 (1.94)

10. Secondary Outcome: Average Pain Assessment in HZ Subjects
Description: as for outcome 9
Time Frame: At Day 90
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 391
Scores on a scale | 0.5 (1.58)

11. Secondary Outcome: Impact of HZ on Quality of Life as Assessed by the Zoster Pain Inventory
Description: PHN persistence refers to pain occurring or persisting between 90-270 days after the rash onset. PHN was assessed via the Zoster Pain Inventory (ZBPI) questionnaire, which includes four pain severity items (worst, least, average, present pain) and seven pain interference items which assess general activity, mood, walking ability, work, relations with others, sleep and enjoyment of life. All of the items are rated on an 11-point Likert scale (0-10). For the severity items, 0 = 'no pain' and 10 = 'pain as bad as you can imagine', whereas for the interference items, 0 = 'does not interfere' and 10 = 'completely interferes'.
Time Frame: At Day 0, 15, 30, 60, 90
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 391
Scores on a scale
  Day 0 | 3.478 (2.707)
  Day 15 | 2.742 (2.749)
  Day 30 | 1.823 (2.459)
  Day 60 | 1.026 (1.931)
  Day 90 | 0.578 (1.471)

12. Secondary Outcome: Impact of HZ on Quality of Life as Assessed by the EuroQoL-Five Digits
Description: EuroQoL-Five Digits (EQ-5D) is a standardised instrument for use as a measure of health outcome and is designed for self-completion by respondents. Its current format is 3-level and 5 dimensional (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The EQ-5D index was derived from the ratings recorded every 3 months for each of the five individual items (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The EQ-5D index/scale goes from 0 (worst health state) to 1 (perfect health state).
Time Frame: At Day 0, 15, 30, 60, 90
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 391
Scores on a scale
  Day 0 | 0.748 (0.207)
  Day 15 | 0.801 (0.198)
  Day 30 | 0.849 (0.207)
  Day 60 | 0.901 (0.175)
  Day 90 | 0.935 (0.140)

13. Secondary Outcome: PHN Direct Medical Costs, Direct Non-medical Costs and Indirect Costs by Payer/Societal Perspective
Description: as for outcome 8
Time Frame: Between Day 90 and Day 270
Population: The analysis was performed on the PHN subjects from the According-To-Protocol cohort (ATP) which included all evaluable patients (i.e. those who met all eligibility criteria and complied with the study procedures defined in the protocol).
Measure: Mean (Standard Deviation); unit: Euro
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 40
Euro
  PHN, Payer | 176 (179)
  PHN, Societal | 426 (663)

14. Secondary Outcome: Worst Pain Assessment in PHN Subjects
Description: as for outcome 9
Time Frame: At Day 90
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 40
Scores on a scale | 5.7 (1.96)

15. Secondary Outcome: Average Pain Assessment in PHN Subjects
Description: as for outcome 9
Time Frame: At Day 90
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 40
Scores on a scale | 4.2 (2.46)

16. Secondary Outcome: Impact of PHN on Quality of Life as Assessed by the Zoster Pain Inventory
Description: as for outcome 11
Time Frame: At Day 0, 15, 30, 60, 90
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 40
Scores on a scale
  Day 0 | 5.967 (2.550)
  Day15 | 6.062 (2.385)
  Day 30 | 5.553 (2.600)
  Day 60 | 4.315 (2.550)
  Day 90 | 3.671 (2.145)

17. Secondary Outcome: Impact of PHN on Quality of Life as Assessed by the EuroQoL-Five Digits
Description: EuroQoL-Five Digits (EQ-5D) is a standardised instrument for use as a measure of health outcome and is designed for self-completion by respondents. Its current format is 3-level and 5 dimensional (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The EQ-5D index was derived from the ratings recorded every 3 months for each of the five individual items (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). The EQ-5D index was 0 (worst health state) to 1 (best health state).
Time Frame: At Day 0, 15, 30, 60, 90
Population: The analysis was performed on the According-To-Protocol cohort (ATP) which included all evaluable patients (i.e. those who mett all eligibility criteria and complied with the study procedures defined in the protocol).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Herpes Zoster Group
Number analyzed (Participants) | 40
Scores on a scale
  Day 0 | 0.592 (0.227)
  Day 15 | 0.582 (0.284)
  Day 30 | 0.542 (0.317)
  Day 60 | 0.688 (0.275)
  Day 90 | 0.732 (0.202)

ADVERSE EVENTS:
Time Frame: Not applicable as serious and other adverse events were not monitored in this study
Description: Serious and other adverse events were not monitored in this study as this a non-interventional study based on pre-existing medical records obtained from a network of general practitioners.There was no assessment of AEs related to any treatment or vaccination in this study, as only burden of Herpes Zoster disease was assessed. Complications and clinical information of HZ cases presented in outcome measures 5-7 and deaths reported in participant flow are obtained from pre-existing medical records.
Arm/Group | Herpes Zoster Group
All-Cause Mortality (participants affected / at risk) | 1/394
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.